CLINICAL TRIAL: NCT00250211
Title: Multimodality Functional Imaging (MRS and Tumor Perfusion) Predicts Tumor Migration, Invasiveness, and Patterns of Failure of Human Glioblastoma Treated With Concurrent Radiation Therapy and Temozolomide
Brief Title: Magnetic Resonance Spectroscopic Imaging (MRS) and Tumor Perfusion of Human Glioblastoma Treated With Concurrent Radiation Therapy and Temozolomide
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Cross Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNS-09-0027 / ethics 21780
Record Dates: First submitted 2005-11-04; First posted 2005-11-08 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2011-10

CONDITIONS: Glioblastoma; Glioma
Keywords: magnetic resonance imaging, functional; radiation therapy; temozolomide; functional imaging; concurrent chemoradiation
MeSH Terms: conditions — Glioblastoma; Glioma | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Functional MRI imaging and tomotherapy

SUMMARY:
The purpose of this study is to learn whether 3 tesla (3T) MRI functional imaging will map a tumor more accurately allowing a more targeted delivery of radiation. The investigators hope to learn whether tomotherapy will be able to deliver higher radiation doses safely to the tumor while sparing the surrounding normal tissue.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed glioblastoma multiforme
* Ages 18-65
* Karnofsky Performance Scale (KPS) equal to or less than 70
* Minimal neurological deficit
* Eligible for concurrent temozolomide chemotherapy

Exclusion Criteria:

* Prior radiation therapy to hand or neck area, chemotherapy, or radiosensitizer

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2005-03; Primary Completion 2011-03 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
determine tumor response and pattern of failure using functional MRI imaging | Study completion
time to disease progression | Study completion

SECONDARY OUTCOMES:
distinguish residual tumor from treatment-related necrosis | study completion
survival
acute late toxicity of tomotherapy and hypofractionation

CONTACTS AND LOCATIONS:
Overall Officials: Bassam Abdulkarim, MD, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada